CLINICAL TRIAL: NCT00644267
Title: Using a Telemedicine System to Promote Patient Care Among Underserved Individuals
Acronym: AHRQ
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Temple University (Other)
Responsible Party: Alfred A. Bove, MD, PhD, Temple University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AHRQ (DHHS)-1R18HS017202; AHRQ-1R18HS017202
Record Dates: First submitted 2008-03-24; First posted 2008-03-26 (Estimated); Last update posted 2010-10-01 (Estimated); Status verified 2010-09

CONDITIONS: Hypertension
Keywords: hypertension; cardiovascular risk; risk score
MeSH Terms: conditions — Hypertension | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Subjects will use a telemedicine system for blood pressure control
  Interventions: Behavioral: Telemedicine
- 2 (No Intervention): Patients with hypertension receiving usual care by a primary care physician
  Interventions: Behavioral: Telemedicine

INTERVENTIONS:
Behavioral: Telemedicine — Telemedicine reporting of blood pressure, weight, physical activity
  Other Names: Internet, world wide web

SUMMARY:
We have established a Telemedicine System for chronic disease management. Based on a personal health record, we have successfully used this system in diverse populations, in over 600 patients, and in multiple disease states (heart failure, CVD risk reduction, gestational diabetes). In this proposal, we will enhance this Telemedicine system to support patient centered care (PCC) by increasing access, incorporating hypertension treatment guideline, quality measures, automating reminders and feedback for both patients and health care providers.

Inner-city, primarily African-American patients (N=252) with uncontrolled hypertension (BP<140/90 mmHg) and who are followed by primary care physicians will be randomized to either a usual care or a telemedicine group (Telemedicine plus usual care). Blood pressure, weight, BMI, blood glucose and lipids, and physical activity will be measured at baseline and at 6 months. We hypothesize that more subjects in the telemedicine group will achieve goal blood pressure than in the control group. This will occur through increases in knowledge, self-management, shared decision-making, and improved doctor-patient interaction. Primary end- point will be the proportion of subjects who achieve goal blood pressure. Secondary end-points will include:

Rate of self-monitoring, steps per day, weight, CVD knowledge, number of patients at medication guidelines, and increased satisfaction with practice. Telemedicine utilization will also be determined. We believe that telemedicine can facilitate PCC and reduce blood pressure in a cost effective manner.

DETAILED DESCRIPTION:
Basic demographic information will be obtained for each subject. The subject's primary care physician's name, contact information, and specialty will be recorded.

All patients will have an initial medical history, physical examination, electrocardiogram, blood studies, urinalysis, height, weight, and blood pressure measurement. Blood pressure measurements will be obtained in the left arm of seated participants after 5 minutes of quiet rest. A minimum of 3 BP readings will be taken. Systolic and diastolic BP will be recorded. Waist circumference will be measured to the nearest 1 cm at the level of the iliac crest while the subject is standing at minimal respiration. A fasting blood sample will be obtained to determine serum cholesterol, LDL, HDL, triglycerides, creatinine, and glucose levels. All participants will receive their values together with a brochure regarding life-style modification (weight loss, smoking cessation, increased physical activity etc as appropriate). The subjects will take a cardiovascular knowledge questionnaire and the CAHPS® Clinician & Group Survey (CAHPS 2006).

Control Patients. Management of the patient's medical condition will be done by the patient's primary care physician. No restriction will be placed on patient care or the number of office visits with their physician(s). If a subject does not have a primary care physician, we will arrange for the subject to be followed in a Temple based primary care practice. At the final visit at 6 months, the control patients will be given the opportunity to be followed by the telemedicine system.

Computer Training: Patients randomized to the telemedicine group will be trained on use of a computer and the Internet and on how to access the Internet and web-site. Each patient will be instructed on the details of Telemedicine system on a demonstration terminal in the research center. At that time, the patient will be provided with login name and password to gain access to the secure telemedicine site. The patient will make data entries with coaching by the research team.

An important feature of the Telemedicine system will be telephone-based data entry and communication. This will be added to the current Internet-based system using an Interactive Voice Recognition (IVR) system, which will enable information transmitted via telephone or Internet to be collected in the central database. Training on use of the IVR system (i.e., how to respond to prompts) will be incorporated into the patient training program for the Internet.

The study patients randomized to the telemedicine group will be given a sphygmomanometer with memory, a scale if needed, and a pedometer to count their steps per day. The participants will receive instructions regarding proper use of these devices. Initially, the subjects will wear a pedometer for 7 consecutive days and record the total number of steps taken each day to obtain their baseline physical activity level. The participants will be given recommendations for a gradual progression toward 10,000 steps/day. Ten thousand steps per day are consistent with approximately 5 miles of walking per day. All participants will be given a logbook and encouraged to record their measurements at least once a week (i.e., blood pressure, weight, average number of steps) over the course of the study. Life style changes, increased exercise and weight loss, can make a significant impact on blood pressure; a weight loss of as little as 10 lbs can reduce blood pressure.

Patients in the telemedicine group will also be provided with a toll-free number with which to access the IVR system (a separate toll-free number will be provided to Hispanic patients for a Spanish language IVR system). This system can be used as an alternate to the web-based data entry screens available to all patients in the Internet arm. Basically, the patient will dial the 800 number and a voice message will ask for the patient ID and password (character strings entered via telephone keypad or spoken in sequence). The numerical values for blood pressure, steps, weight, and cigarettes smoked can be entered via voice recognition or by the keypad. Voice messages from the patient will also be permitted. These will be spoken after a prompt, and will be designed to provide a short (i.e. 1 minute) voice transmission that will be stored as a voice file (WAV) to the telemedicine system database. Data entered via the IVR system will be inserted into the patient's personal health record stored in the Telemedicine database.

ELIGIBILITY:
Inclusion Criteria:

* uncontrolled hypertension
* systolic blood pressure > 140
* access to a telephone or internet

Exclusion Criteria:

* angina
* cognitive defects, dementia
* end stage renal disease
* living in nursing or boarding homes
* pregnant
* unable to sign informed consent
* unable to use a scale, sphygmomanometer, pedometer

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2008-04; Primary Completion 2010-10 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
Lowering of blood pressure from hypertension to prehypertension in 50% of study subjects | 6 months

SECONDARY OUTCOMES:
significant reduction in systolic blood pressure in the telemedicine arm | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Alfred A Bove, MD PhD, Principal Investigator — Temple University
Locations (1):
- Temple University School of Medicine, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Bove AA, Homko CJ, Santamore WP, Kashem M, Kerper M, Elliott DJ. Managing hypertension in urban underserved subjects using telemedicine--a clinical trial. Am Heart J. 2013 Apr;165(4):615-21. doi: 10.1016/j.ahj.2013.01.004. Epub 2013 Mar 6. PMID 23537980